CLINICAL TRIAL: NCT04684719
Title: Type O Whole Blood and Assessment of Age During Prehospital Resuscitation (TOWAR) Trial
Brief Title: Type O Whole Blood and Assessment of Age During Prehospital Resuscitation Trial
Acronym: TOWAR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jason Sperry (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Jason Sperry, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY20110430; W81XWH-16-D-0024 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2020-12-18; First posted 2020-12-24 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Hemorrhagic Shock; Traumatic Injury
Keywords: hemorrhage; trauma; whole blood
MeSH Terms: conditions — Shock, Hemorrhagic; Wounds and Injuries; Hemorrhage | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Whole Blood (Experimental): Subjects will receive up to two units of whole blood as collected by local blood bank procedures and stored at 1-6 degrees Celsius initiated in the prehospital phase of care.
  Interventions: Biological: low titer whole blood
- Standard Care (Active Comparator): Subjects will receive prehospital crystalloid infusion or blood component transfusion resuscitation per site standard care for the respective Emergency Medical unit/service.
  Interventions: Biological: Standard Care

INTERVENTIONS:
Biological: low titer whole blood — low titer whole blood, group O kept to either 21 days or 35 days based upon which preservation process is employed at each respective participating site
  Arms: Whole Blood
Biological: Standard Care — crystalloid infusion or blood component transfusion resuscitation
  Arms: Standard Care

SUMMARY:
Open label, multi-center, pre-hospital randomized trial utilizing 10 level-1 trauma centers designed to determine the efficacy and safety of low titer whole blood resuscitation as compared to standard of care resuscitation in patients at risk of hemorrhagic shock and to appropriately characterize the hemostatic competency of whole blood relative to its age.

ELIGIBILITY:
Inclusion Criteria:

1.) Injured patients at risk of hemorrhagic shock being transported from scene or referral hospital to a participating TOWAR trial site that meet requirements for initiation of blood or blood component transfusion

AND

2A.) Systolic blood pressure ≤ 90mmHg and tachycardia (HR ≥ 108) at scene, at outside hospital or during transport OR

2B.) Systolic blood pressure ≤ 70mmHg at scene, at outside hospital or during transport

Exclusion Criteria:

1. Wearing NO TOWAR opt-out bracelet
2. Age > 90 or < 18 years of age
3. Isolated fall from standing injury mechanism
4. Known prisoner or known pregnancy
5. Traumatic arrest with > 5 minutes of CPR without return of vital signs
6. Brain matter exposed or penetrating brain injury (GSW)
7. Isolated drowning or hanging victims
8. Objection to study voiced by subject or family member at the scene
9. Inability to obtain IV or intraosseous access
10. Isolated burns without evidence of traumatic injury

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1020 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2025-07-28 (Actual); Study Completion 2025-08-12 (Actual)

PRIMARY OUTCOMES:
30-day mortality | Enrollment through 30 days
  All cause mortality within 30 days

SECONDARY OUTCOMES:
Age of whole blood | During Procedure
  Age of units of whole blood in days categorized into young (1-14 days) and old (>14 days) and compared across primary and secondary outcomes
3-hour mortality | Enrollment through 3 hours
  Death within 3 hours of enrollment
6-hour mortality | Enrollment through 6 hours
  Death within 6 hours of enrollment
24-hour mortality | Enrollment through 24 hours
  Death within 24 hours of enrollment
In-hospital mortality | Enrollment through hospital discharge or 30 days
  Death prior to hospital discharge
Time to death | Enrollment through death or 30 days
  Time in days from enrollment to death
Blood and blood component transfusion type | Enrollment through 24 hours
  Type of blood or blood component required for transfusion
Blood and blood component transfusion amount | Enrollment through 24 hours
  Number of units of blood or blood component transfused
Time to blood and blood component transfusion | Enrollment time to first transfusion
  Amount of time from enrollment to transfusion of blood or blood component
Multiple Organ Failure (MOF) | Enrollment through 7 days or ICU discharge
  Organ dysfunction will be evaluated via the Denver Post-injury Multiple Organ Failure Score. Patients who are never admitted to the Intensive Care Unit (ICU) or those with a length of ICU stay of less than 48 hours will be considered to have a Denver score of 0. A summary of the Denver score may be calculated by summing the worst scores of each of the individual systems over the course of the ICU stay. A summary Denver score > 3 will be classified as MOF.
Hospital-acquired pneumonia | Number of participants who develop pneumonia through 30 days
  Pneumonia acquired during hospitalization per Center for Disease Control (CDC) criteria
blood stream infection | Number of participants who develop blood stream infection through 30 days
  Blood stream infection during hospitalization per CDC criteria
Acute Respiratory Distress Syndrome (ARDS) | Number of participants who develop ARDS through 30 days
  The Berlin definition for mild ARDS (PaO2/FIO2, ≤ 300 mm Hg + timing, imaging and origin criteria) will be utilized as a threshold value to determine the incidence of ARDS and will be further stratified into Moderate (PaO2/FIO2, ≤ 200 mm Hg) and Severe (PaO2/FIO2, ≤ 100 mm Hg).
Prothrombin Time (PT) | Enrollment through 60 minutes and 24 hours
  Measurement of platelet hemostatic function
International Normalized Ratio (INR) | Enrollment through 60 minutes and 24 hours
  Measurement of platelet hemostatic function
Incidence of coagulopathy by rapid thrombelastography (rTEG) | Enrollment through 60 minutes and 24 hours
  Coagulopathy as indicated by rTEG measures
rTEG platelet function | Enrollment through 60 minutes and 24 hours
  rTEG measurement of platelet hemostatic function
Time to hemostasis | Enrollment through 4 hours
  Ability to reach nadir transfusion requirement of 1 unit of red blood cells in a 60-minute time period in the first 4 hours following arrival
Transfusion reaction | Enrollment through 24 hours
  Any transfusion complication
whole blood aggregometry | Enrollment through 60 minutes
  platelet function test using low-dose collagen as a stimulus

CONTACTS AND LOCATIONS:
Overall Officials: Jason L Sperry, MD, Principal Investigator — University of Pittsburgh
Locations (10):
- United States (10):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Louisville, Louisville, Kentucky
  - University of Mississippi Medical Center (UMMC), Jackson, Mississippi
  - University of Cincinatti, Cincinnati, Ohio
  - Metrohealth Systems, Cleveland, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Health Science Center at Houston, Houston, Texas
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
De-identified data may be shared with the funding agency as well as other researchers upon request to the Principal Investigator.
Supporting Information: Study Protocol, ICF
Time Frame: Data will become available after publication of the primary manuscript.
Access Criteria: Requests for data will be submitted in writing and reviewed by the Principal Investigator.

REFERENCES:
- [Derived] Brunskill SJ, Disegna A, Wong H, Fabes J, Desborough MJ, Doree C, Davenport R, Curry N, Stanworth SJ. Blood transfusion strategies for major bleeding in trauma. Cochrane Database Syst Rev. 2025 Apr 24;4(4):CD012635. doi: 10.1002/14651858.CD012635.pub2. PMID 40271704
- [Derived] Meizoso JP, Cotton BA, Lawless RA, Kodadek LM, Lynde JM, Russell N, Gaspich J, Maung A, Anderson C, Reynolds JM, Haines KL, Kasotakis G, Freeman JJ. Whole blood resuscitation for injured patients requiring transfusion: A systematic review, meta-analysis, and practice management guideline from the Eastern Association for the Surgery of Trauma. J Trauma Acute Care Surg. 2024 Sep 1;97(3):460-470. doi: 10.1097/TA.0000000000004327. Epub 2024 Mar 27. PMID 38531812

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-23): https://cdn.clinicaltrials.gov/large-docs/19/NCT04684719/Prot_SAP_000.pdf
  • Informed Consent Form (2024-10-18): https://cdn.clinicaltrials.gov/large-docs/19/NCT04684719/ICF_001.pdf